CLINICAL TRIAL: NCT04820621
Title: Investigation of the Pharmacokinetics, Safety and Tolerability of Runcaciguat in Participants With Hepatic Impairment (Classified as Child Pugh A or B) and in a Control Group of Age-, Weight-, and Gender-matched Participants Following a Single Oral 15 mg Modified Release (MR) Tablet Dose in a Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: Study of the Influence of Liver Function on Blood Concentrations of Runcaciguat in Participants With Different Degrees of Liver Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study is prematurely terminated due to changes in sponsor's overall development strategy. The decision of termination is not related to any safety concern of the compound.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19620; 2020-005716-22 (EudraCT Number)
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — BAY 1101042

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants with mild hepatic impairment (Experimental): All participants will receive a single oral dose in the fasted state on Day 1.
  Interventions: Drug: Runcaciguat (BAY1101042)
- Participants with moderate hepatic impairment (Experimental): All participants will receive a single oral dose in the fasted state on Day 1.
  Interventions: Drug: Runcaciguat (BAY1101042)
- Participants with normal hepatic function (Experimental): All participants will receive a single oral dose in the fasted state on Day 1.
  Interventions: Drug: Runcaciguat (BAY1101042)

INTERVENTIONS:
Drug: Runcaciguat (BAY1101042) — Given as 1 x 15 mg modified release [MR] tablet

SUMMARY:
Researchers are looking for a better way to treat people with chronic kidney diseases. Before a treatment can be approved for patients to take, researchers do clinical studies to better understand its safety and what happens to the drug in the body.

In this study researchers will investigate how the liver function influences blood concentrations of runcaciguat in participants with different degrees of liver impairment compared to participants with normal liver function.

The participants will all take one tablet with 15 mg runcaciguat by mouth. Prior to inclusion into the study, all participants will have a screening examination within 21 to 2 days prior to dosing to check eligibility for study participation.

During the study, all of the participants will stay at the study site for up to 8 days (from Day -1 to Day 7), whereby Day 6 and 7 might also be performed in an ambulatory setting. Blood and urine samples will be collected. The physician will check the participants' heart health using an electrocardiogram (ECG) and by measuring blood pressure and heart rate. The participants will answer questions about their wellbeing and taken medications.

The participants will have a follow-up examination 7 to 11 days after dosing to follow-up their health.

Each participant will be in the study for approximately 5 weeks. The entire study will last about 9 months.

ELIGIBILITY:
Inclusion Criteria:

Age

* Participant must be 18 to 79 years of age (inclusive) at the time of signing the informed consent.

Weight

* Body mass index (BMI) within the range 18 to 35 kg/m^2 (inclusive). Sex and Contraceptive/Barrier Requirements
* Male and female white participants. Main Inclusion Criteria for participants with hepatic impairment
* Participants with hepatic impairment (Child Pugh A or B).
* Participants with stable liver disease in the last 2 months. Main Inclusion Criteria for control group of participants
* Healthy male and female white participants.
* Mean age and body weight in the control group and in the two groups with hepatic impairment (Child Pugh A and B) should not vary by more than ±10 years and ±10 kg.
* Gender-matched.

Exclusion Criteria:

Main exclusion Criteria for all participants Medical and surgical history

* Participants with a medical disorder, condition, or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator or the sponsor.

Medication, drug use and special behavioral patterns

* Suspicion of drug or alcohol abuse. Other
* Participation in another clinical trial within 3 months (for previous multi-dose study) or 1 month (for previous single dose study) before dosing.
* Exclusion periods from other studies or simultaneous participation in other clinical studies.

coronavirus disease 2019 (COVID-19) specific exclusion criteria

* History of COVID-19.
* Contact with severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) positive or COVID-19 patient within the last 4 weeks prior to admission to the clinical unit
* Positive SARS-CoV-2 viral polymerase chain reaction (PCR) test

Main exclusion Criteria for participants with hepatic impairment Medical and surgical history

* Pre-existing diseases beside hepatic impairment for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Evidence of hepatic encephalopathy related to chronic liver disease > grade 2 (exclusion by Number Connection Test).
* Congestive heart failure of New York Heart Association grade III or IV.
* History of conspicuous bleeding within the past 3 months.
* Severe arrhythmia requiring antiarrhythmic treatment within the past 3 months.
* Participants with diabetes mellitus with a glycohemoglobin A1c (HbA1c) >9%.
* Severe ascites of more than 6 L (estimated by ultrasound).
* Participants with primary and secondary biliary cirrhosis.
* Participants with sclerosing cholangitis. Electrocardiogramm (ECG), blood pressure, heart rate
* Systolic blood pressure below 100 mmHg or above 169 mmHg.
* Diastolic blood pressure below 50 and above 95 mmHg.
* Resting heart rate below 50 beats per minute (bpm) or above 95 bpm. Laboratory examination
* Platelet count < 40 x 10^9/L.
* Hemoglobin <9 g/dL.
* Alkaline phosphatase (AP) ≥ 4 times the upper limit of normal (ULN).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) in conjunction with gamma glutamyl transpeptidase (GGT) ≥4 times the ULN (an isolated elevation of GGT above 4 times ULN will not exclude the participant).
* Serum albumin <20 g/L.
* Prothrombin time (Quick test) <40%.
* Renal failure with an estimated glomerular filtration rate (eGFR) ≤ 40 mL/min/1.73 m^2 (according to CKD-EPI equation).

Main Exclusion criteria for control group of participants Medical and surgical history

* A history of relevant diseases of vital organs, the central nervous system, or other organs.
* Liver insufficiency or active liver disease, which may include unexplained persistent transaminase elevations.
* Renal impairment with an estimated glomerular filtration rate (eGFR) ≤80 mL/min/1.73 m^2 (according to CKD-EPI equation).
* Known or suspected liver disorders (e.g. Morbus Gilbert/Meulengracht) and bile secretion/flow (cholestasis, also history of it).

Medication, drug use and special behavioral patterns

* Regular use of therapeutic or recreational drugs, e.g. carnitin products, anabolics, high dose vitamins.

Laboratory examination

* Relevant deviation from the normal range in clinical chemistry (including thyroid stimulating hormone [TSH]), hematology, coagulation or urinalysis as judged by the investigator.
* Increase of liver enzymes (e.g. ALT, AST, alkaline phosphatase, gamma glutamyl transpeptidase or total bilirubin) above ULN.
* Increase of lipase and amylase (despite isolated marginal increases of lipase or amylase to account for variability of the parameters, and the participant is asymptomatic and has no other laboratory changes assuming disease based on medical judgment).
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus (HIV) antibodies 1+2/HIV p24 antigen (HIV-1/2 combi test).

Electrocardiogramm (ECG), blood pressure heart rate

* Systolic blood pressure below 100 or above 145 mmHg at screening.
* Diastolic blood pressure below 50 or above 95 mmHg at screening.
* Resting heart rate below 50 or above 95 bpm at screening.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve from zero to infinity after single (first) dose (AUC) of BAY1001042 | From dosing day (Day 1) up to 12 days post dose
  AUC(0-tlast) will be used as main parameters if mean AUC(tlast - ∞) >20% of AUC
Unbound AUC (AUCu) of BAY1001042 | From dosing day (Day 1) up to 12 days post dose
  AUC(0-tlast)u will be used as main parameters if mean AUC(tlast - ∞) >20% of AUC
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of BAY1001042 | From dosing day (Day 1) up to 12 days post dose
Unbound Cmax (Cmax,u) of BAY1001042 | From dosing day (Day 1) up to 12 days post dose

SECONDARY OUTCOMES:
Numbers of participants with treatment-emergent adverse events (TEAEs) and study intervention related TEAE | From start of treatment up to 10 days after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.